CLINICAL TRIAL: NCT03542695
Title: Use of 64Cu-DOTA-Alendronate PET Imaging for Localization and Characterization of Breast Calcifications
Brief Title: 64 Cu-DOTA-alendronate PET Imaging in Localizing and Characterizing Breast Calcifications in Participants Before Undergoing Mastectomy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18112; NCI-2018-00890 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 18112 (Other: City of Hope Medical Center)
Record Dates: First submitted 2018-05-18; First posted 2018-05-31 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Breast Carcinoma; Calcification
MeSH Terms: conditions — Breast Neoplasms; Calcinosis | interventions — Pharmacogenomic Variants; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (64Cu-DOTA-alendronate, PET/CT scan) (Experimental): Participants receive 64Cu-DOTA-alendronate IV and undergo PET/CT imaging 60 minutes after injection. Participants with sufficient levels of residual radioactivity may undergo repeat imaging on day 1 as determined by the study team.
  Interventions: Procedure: Computed Tomography; Drug: Copper Cu-64-DOTA-alendronate; Other: Pharmacokinetic Study; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT; CT SCAN; tomography
Drug: Copper Cu-64-DOTA-alendronate — Given IV
  Other Names: 64Cu-DOTA-alendronate; [64Cu]-DOTA-alendronate
Other: Pharmacokinetic Study — Correlative studies
  Other Names: PHARMACOKINETIC; PK Study
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This early phase I pilot trial studies how well 64Cu-DOTA-alendronate positron emission tomography (PET) imaging work in localizing and characterizing breast calcifications (small calcium deposits) in participants before undergoing mastectomy. Diagnostic procedures, such 64Cu-DOTA-alendronate PET, may detect calcification and help doctors predict cancer associated calcification within breast tissue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the uptake (maximum standardized uptake value [SUVmax]) of 64Cu-DOTA-alendronate in female patients with biopsy-proven malignant breast calcifications.

SECONDARY OBJECTIVES:

I. To compare uptake of 64Cu-DOTA-alendronate on PET -computed tomography (CT) with histology after mastectomy.

OUTLINE: This is a dose-escalation study of 64Cu-DOTA-alendronate.

Participants receive 64Cu-DOTA-alendronate intravenously (IV) and undergo PET/CT imaging 60 minutes after injection. Participants with sufficient levels of residual radioactivity may undergo repeat imaging on day 1 as determined by the study team.

After completion of study , participants are followed up for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of calcifications on mammogram
* Biopsy confirmed malignancy associated calcifications in at least one breast
* Biopsy confirmed benign calcifications in at least one breast (same or contralateral breast)
* Planned total mastectomy for treatment
* Ability to provide informed consent
* Negative serum pregnancy test
* No evidence of impaired hepatic or kidney function

Exclusion Criteria:

* Participants who do not have residual calcifications present on mammogram following biopsy
* Concurrent malignancy other than non-melanoma skin cancer
* Patients with known metastatic disease
* Patients who have received prior treatment for the current breast cancer
* Patients currently using oral bisphosphonate therapy
* Patients with injection of other radioactive material within 90 days
* Inability to provide informed consent
* Pregnant or lactating patients
* Patients with impaired kidney function (creatinine >= 1.3 mg/dL or < 0.6 mg/dL)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Maximum standardized uptake value (SUVmax) of 64Cu-DOTA-alendronate in evaluating tumor size and calcifications | Up to 7 days
  Tumor size sensitivity and the ability to detect calcifications will be compared to the extent of calcifications seen on mammogram.

SECONDARY OUTCOMES:
Uptake of 64Cu-DOTA-alendronate on positron emission tomography (PET) scan compared to histology after mastectomy | Up to 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Jones, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States